CLINICAL TRIAL: NCT02502500
Title: An Open-label Study in Healthy Subjects to Assess the Effect of Once-daily Multiple Dosing of AKB-6548 on the Pharmacokinetics of the CYP2C9 Substrate Celecoxib
Brief Title: Effect of AKB-6548 on the Pharmacokinetics of Celecoxib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AKB-6548-CI-0019
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Celecoxib; vadadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib (Active Comparator): Celecoxib
  Interventions: Drug: Celecoxib
- AKB-6548 and Celecoxib (Experimental): AKB-6548; celecoxib
  Interventions: Drug: Celecoxib; Drug: AKB-6548

INTERVENTIONS:
Drug: Celecoxib
  Other Names: CELEBREX®
Drug: AKB-6548
  Arms: AKB-6548 and Celecoxib

SUMMARY:
To assess the single dose pharmacokinetics (PK) of celecoxib in healthy subjects when administered alone and following multiple daily doses of AKB-6548.

DETAILED DESCRIPTION:
To assess the single dose plasma pharmacokinetics (PK), safety, and tolerability of celecoxib in healthy subjects with CYP2C9 extensive metabolizer (EM) genotype when administered alone and following multiple daily doses of AKB-6548.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 55 years of age, inclusive, and with a body mass index between 18 and 30 kg/sq.meters, inclusive.
* Subjects with the following genotype based upon pharmacogenetic testing results: CYP2C9 EM: *1*1.

Exclusion Criteria:

* Current or past history of cardiovascular, cerebrovascular, pulmonary, renal or liver disease.
* Positive serology results for HBsAg, HCV, and HIV at Screening.
* Significant renal impairment as evidenced by an estimated glomerular filtration rate (eGFR) of <65 mL/minute/1.73 sq.meters.
* Known hypersensitivity to celecoxib or sulfonamides.
* History of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs.
* Known active cancer or history of chemotherapy use within the previous 24 months.
* Current or past history of gastric or duodenal ulcers or other diseases of the GI tract (including gastric bypass surgeries) that could interfere with absorption of study drug.
* Current or past history of gastrointestinal bleeding.
* Any history of alcohol or drug abuse within the previous year prior to Screening.
* Subjects with a known history of smoking and/or have used nicotine or nicotine containing products within the past 6 months.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
PK parameters (Cmax) | pre-dose to 48 hours post-dose
  maximum observed plasma concentration (Cmax) for celecoxib
PK parameters (time to reach Cmax ) | pre-dose to 48 hours post-dose
  time to reach Cmax for celecoxib
PK parameters (t½) | from pre-dose to 48 hours post-dose
  terminal elimination half-life (t½) for celecoxib
PK parameters (AUC0-t) | pre-dose to 48 hours post-dose
  concentration (AUC0-t) for celecoxib
PK parameters (area under the plasma concentration-time curve from 0 to last quantifiable) | pre-dose to 48 hours post-dose
  area under the plasma concentration-time curve from 0 to last quantifiable
PK parameters (AUC0-inf) | from pre-dose to 48 hours post-dose
  AUC from time 0 to infinity (AUC0-inf) for celecoxib
PK parameters (CL/F) | pre-dose to 48 hours post-dose
  apparent oral clearance (CL/F) for celecoxib
PK parameters (Vz/F) | pre-dose to 48 hours post-dose
  apparent volume of distribution during the terminal phase (Vz/F) for celecoxib

SECONDARY OUTCOMES:
Safety and Tolerability will be measured by vital signs | up to ten days
  The safety and tolerability of the single doses of celecoxib alone and in combination with AKB-6548 will be monitored for vital signs, clinical laboratory assays
Safety and Tolerability will be monitoring of adverse events (AEs) | up to ten days
  The safety and tolerability of the single doses of celecoxib alone and in combination with AKB-6548 will be monitored for adverse events (AEs)
Safety and Tolerability will be measured by clinical assays | up to ten days
  The safety and tolerability of the single doses of celecoxib alone and in combination with AKB-6548 will be monitored for clinical laboratory assays

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH

IPD SHARING:
Plan to Share IPD: Undecided